CLINICAL TRIAL: NCT06608706
Title: The Key to Integrated Trauma Treatment in Psychosis (Kit) Trial: a Pragmatic, Multicenter Effectiveness RCT of EMDR for Trauma Symptoms in Schizophrenia Spectrum Disorders
Brief Title: The Key to Integrated Trauma Treatment in Psychosis Trial
Acronym: KIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helgeland Hospital Trust (Other)
Responsible Party: Principal Investigator, Else-Marie Løberg, Principal Investigator (Professor, PhD, Psychologist), Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 714736
Record Dates: First submitted 2024-09-06; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Psychiatric Diagnosis; Schizophrenia Disorders; Psychological Trauma, Historical
Keywords: Psychosis; EMDR; Trauma treatment; Schizophrenia spectrum disorders; Childhood trauma; Psychological trauma; PTSD
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Historical Trauma; Psychotic Disorders; Psychological Trauma; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma-focused therapy: EMDR for psychosis and treatment as usual (TAU) (Experimental): Patients randomized to receive max. 26 sessions of EMDR for psychosis.
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR) for psychosis
- Treatment as usual (TAU) and waiting list (WL) (No Intervention): Patients randomized to continue with treatment as usual (TAU) for 6 months as a waiting list (WL) control group. TAU consists of an individual combination of treatments for SSDs in line with Norwegian national guideline (e.g. medication, cognitive therapy, work training, music therapy).

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing (EMDR) for psychosis — EMDR aims to treat and process trauma by safely retrieving the trauma memories while taxing the working memory. EMDR targets trauma symptoms through memory reprocessing of traumatic memories, and consists of eight flexible phases: history taking/case conceptualization; preparation for memory reprocessing; assessment/identification of a target memory; desensitization/reprocessing; installation of positive cognition; body scan; closure; and re-evaluation. EMDR in the current trial has psychosis-specific adaptations including focus on psychoeducation, preparation for reprocessing and patient safety. Techniques targeting dissociation, psychotic symptoms and psychosis-related challenges are included.
  Arms: Trauma-focused therapy: EMDR for psychosis and treatment as usual (TAU)

SUMMARY:
Schizophrenia spectrum disorders (SSDs) have a significant trauma etiology: trauma has been reported in 65 - 80% in this patient group and have a negative impact on prognosis. Trauma treatment is currently not offered in SSDs due to a lack of evidence. KIT is a pragmatic trial comparing the effectiveness of added trauma focused therapy, Eye Movement Desensitization and Reprocessing (EMDR) to standard treatment in SSDs.

The study will compare EMDR as add on to treatment as usual (TAU) to TAU in patients with schizophrenia spectrum disorders (SSDs). The overall aim is to examine the effectiveness of EMDR on trauma symptoms in SSDs.

Participants will receive max. 26 sessions of EMDR, and complete assessments before, during and after the course of therapy, in addition to a period of time (6 months) after therapy to examine long-term effects.

DETAILED DESCRIPTION:
The KIT trial is a pragmatic, assessor-blinded, parallel 2-group, superiority randomized trial comparing the addition of EMDR to treatment as usual (TAU) versus waiting list (WL) and TAU for EMDR on symptoms of trauma in patients with SSDs. Participants will be randomized (1:1, block randomization by center and gender) to one of the two groups.

Aims, hypotheses, objectives:

* The primary aim is to investigate the effectiveness of EMDR as an add-on treatment for SSDs in standard clinical practice to target trauma symptoms.
* The secondary aim is to improve personalized therapy through the exploration of clinical stratification variables that may influence the effectiveness of EMDR.
* The long-term aim is to guide clinical practice and, if shown to be effective, to implement EMDR for patients with SSDs.
* The primary objective: EMDR and treatment as usual (TAU) compared to waiting list (WL) and TAU will reduce symptoms of trauma as measured by the ITQ (the International Trauma Questionnaire) in SSDs.
* The secondary objective: Stratification variables (trauma profile e.g. type, severity, timing; gender; biomarkers of stress and immune system reactivity; digital biomarkers of autonomous stress reactivity) influence the effectiveness of EMDR.

Expected results during the project period:

* The EMDR group will show less trauma symptoms compared to the WL control group by the end of treatment and possibly better functioning.
* No differences for costs nor serious adverse events will emerge between the groups at the end of treatment.
* Better outcomes are expected for trauma characterized by mild to moderate severity and later onset (e.g. related to experience of psychosis) as compared to CT (e.g. abuse and neglect).
* Although exploratory, patients with high levels of inflammation markers and/or hyperarousal and autonomous reactivity to trauma benefit most from EMDR.

EMDR for psychosis therapists: Eighteen trial therapists are currently fully trained in EMDR for psychosis in collaboration with Dr. Varese and colleagues at Manchester University, and receive monthly supervision. At least 24 more will be trained by early 2025. Assuming some therapist drop-out, 40 trial therapists will be recruiting SSD patients from their patient lists.

Assessments: Assessments will be performed for both groups by blinded research personnel at baseline, mid-treatment (12 weeks), end of treatment (6 months), 6- and 12-months post randomisation after end of treatment, in addition to digital patient feedback every 2 weeks from baseline to end of treatment at 6 months. The follow-up period after end of treatment is to examine long-term effects.

Eligible participants will be given initial information (verbal, web page, pamphlets) by the trial therapists, and then verbal and written information by research staff and asked for informed consent to partake in the trial. Primary outcome will be measured by the ITQ, a validated measure assessing reliable and clinically significant treatment-related change in trauma symptoms, including symptoms of PTSD and complex PTSD, used in outpatient clinics in Norway. Demographic and clinical information will be supplemented by clinical records and national health registers (e.g. Legemiddel-registeret, Kontroll og utbetaling av helserefusjoner, Kommunalt pasient og bruker-register, Norsk pasientregister, Nasjonalt kvalitetsregister for behandling i psykisk for voksne). Healthcare costs (e.g. use of all health care, health related financial support, transportation) will be captured by the study nurses at each assessment point and through health registers.

Patients' experience of trauma symptoms, working alliance and recovery will be assessed through Norse Feedback digital self-report. The digital assessment of the main outcome trauma symptoms (ITQ) will be captured every 2 weeks to closely monitor symptom fluctuations, while recovery and therapist alliance follow the time points of the study nurse assessments. This decentralised assessment is deemed particularly suitable in mental health. Assessment of somatic status (heartrate, weight, blood pressure) will be supplemented by blood samples of inflammation markers (CRP, IL6 and S-cortisol) and blood samples to the Bergen Psychosis Biobank for later analysis (e.g. IL18). The digital biomarkers heart rate variability, respiration rate (electro- cardiography/photoplethysmography), activation/ movement (actigraphy) and skin conductance (electrodermal activity) will be measured in-session by BioPoint wristworn biosensor. Trial therapists will rate fidelity, patient safety related adverse events (AE) and symptom exacerbation after each session, and variables facilitating implementation before/after trial participation. For symptom-specific items on suicidality, psychosis, substance abuse and hospitalisations. A sub-group of 30 patients will be asked about their experience of the therapy with a qualitative interview after treatment.

Work packages: Quality of assessments and analysis will be ensured by organising themes in work packages (WP) headed by national experts; WP0 Study management, WP1 Clinical outcome, WP2 Somatic status and biomarkers, WP3 Trauma characteristics, WP4 Treatment alliance and user experience, WP5 Study imple-mentation, WP6 Health economic evaluation.

Protocol adherence: Hospital Clinical Monitor will ensure protocol implementation and site responsibility. The protocol will be adhered to by all trial personnel, including trial therapists and local PIs to ensure patient safety and trial quality. There will be frequent meetings across sites and written agreements on site responsibility. All sites will use electronic report files (CRF) via Viedoc for patient case report forms.

Organization: The KIT trial is organized in Bergen Psychosis Research Group (BPRG) at Haukeland University Hospital. BPRG has extensive experience from clinical trials on SSDs (ClinicalTrials.gov IDs NCT00932529, NCT01446328, NCT03340909, NCT02597439, NCT02146547).

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 16 years
2. diagnosis of F20-29 in the ICD-10 assessed using SCID 5 CV
3. reporting trauma > 1 month prior to assessment
4. being currently distressed by the reported trauma(s), i.e., ≥ 5 (from 0 = not at all, to 10 = extremely) on item 21c on the Trauma and Life Events Checklist (TALE)
5. able and motivated for engaging in trauma focused (TF) therapy
6. able to understand and give informed consent; consent capacity for psychological treatment choices and consent to study procedures.

Exclusion Criteria:

1. primary diagnosis of substance use/alcohol dependence
2. inability to understand spoken Norwegian
3. organic psychosis or a neurological disorder
4. acute state of psychosis defined as:

   1. hospitalized in an acute ward the last 6 weeks or
   2. major change in antipsychotic medication type or started/stopped antipsychotic medication last 6 weeks or
   3. other mental health crises last 6 weeks
5. current or previous (past 6 months) TF therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Trauma symptoms | From baseline to end of treatment at 6 months.
  Primary outcome is trauma symptoms as measured by the International Trauma Questionnaire. PTSD symptom scale range from 0 to 24. Higher scores indicate more sever trauma symptoms.

SECONDARY OUTCOMES:
Severity of psychosis symptoms | From baseline to end of treatment at 6 months.
  Secondary outcome is psychosis symptoms as measured by the The Positive and Negative Syndrome Scale (PANSS), which ranges from 30 to 210, with higher scores indicating more severity.
The rate of autonomic arousal during trauma processing | Baseline to end of treatment at 6 months.
  Digital biomarkers measured with BioPoint wrist-worn device. Physiological stress reactivity is recorded non-invasively and continuously, offering an especially suitable means for monitoring objective physiological responses. Real-time assessments of hyperarousal, autonomic and somatic reactivity, and stress reactivity (including heart rate variability, skin conductance, respiration, and actigraphy) will be administered during EMDR sessions.
Inflammation | Baseline and end of treatment at 6 months
  Measure of inflammation markers (CRP, IL6) using blood samples

OTHER OUTCOMES:
Clinical stratification by trauma type and severity measured by the Childhood Trauma Questionnaire | Baseline to end of treatment at 6 months.
  Trauma type and severity as measured by the Childhood Trauma Questionnaire short form (CTQ-SF). CTQ-SF ranges from 25 to 125, with higher scores indicating more severe childhood trauma. Subscale scores range from 5-25 for the following sub scales: physical, emotional and sexual abuse, and physical and emotional neglect.
Adverse events | Baseline to end of treatment at 6 months.
  No differences in adverse events is expected between the groups.
Health care costs | Baseline to end of treatment at 6 months.
  No difference in health care costs is expected between the groups.
Clinical stratification by trauma type and severity measured by the Traumatic experiences checklist | Baseline to end of treatment at 6 months.
  Severity and type of trauma measured by the Traumatic Experiences Checklist (TEC). The TEC indicates the presence of trauma on a scale from 0-29, higher scores indicating more exposure. TEC also include composite scores from 0-12 by developmental period, where higher scores indicate more severity.
Clinical stratification by trauma symptoms measured by the International Trauma Questionnaire | Baseline to end of treatment at 6 months.
  Trauma symptoms measured by the International Trauma Questionnaire (ITQ). The ITQ ranges from 0-24 for PTSD symptoms and 0-24 for symptoms of complex PTSD, where higher scores indicate more severe symptoms. There is also a diagnostic algorithm for PTSD and complex PTSD status.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Helgeland Hospital HF, Sandnessjøen

IPD SHARING:
Plan to Share IPD: No
This is not feasible due to Norwegian policies in clinical research.

REFERENCES:
- See also: Trial web-page — https://www.helse-bergen.no/avdelinger/psykisk-helsevern/forskingsavdelinga-divisjon-psykisk-helsevern/kit-trial/